CLINICAL TRIAL: NCT04052243
Title: An International Multicenter Observational Study to Assess the Hemodynamic Effects of Balloon Pulmonary Angioplasty (BPA) at Rest and During Exercise in Chronic Thromboembolic Pulmonary Hypertension (CTEPH) or Chronic Thromboembolic Pulmonary Disease (CTED) Patients (EXPERT-BPA)
Brief Title: Hemodynamic Effects of BPA at Rest and During Exercise in CTEPH
Acronym: EXPERT-BPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Nagoya University (Other); Department of Pulmonary Circulation and Thromboembolic Diseases, Medical Center for Postgraduate Med (Other)
Responsible Party: Principal Investigator, Mads Jønsson Andersen, Principal Investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EXPERT-BPA
Record Dates: First submitted 2019-07-11; First posted 2019-08-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: Exercise is added to the resting right heart catheterization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Exercise is added to resting right heart catheterization
  Interventions: Diagnostic Test: Invasive exercise testing

INTERVENTIONS:
Diagnostic Test: Invasive exercise testing — Invasive hemodynamic exercise testing

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is characterized by obstruction of the pulmonary vasculature by residual organized thrombi, leading to increased pulmonary vascular resistance (PVR), progressive pulmonary hypertension, and right heart failure.

Medical therapy and balloon angioplasty (BPA) are effective treatment alternatives in lowering pulmonary pressures and increasing pulmonary flow.

The aim of this study is to assess the hemodynamic effects of BPA or medical therapy on the pressure-flow relationship in the pulmonary vasculature and the pulmonary vascular compliance.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension [CTEPH] is a rare condition with a significant risk of morbidity and mortality. The primary cause of CTEPH is thrombotic lesions, which did not resolve after acute pulmonary embolism. This causes increased pulmonary vascular resistance [PVR], leading to secondary remodeling of pulmonary arteries causing pulmonary hypertension and ultimately progressive right heart failure. The treatment of choice is surgical pulmonary endarterectomy [PEA], however up to 40% cases are not treated surgically, due to operability, anatomic location of the lesions, patient choice and comorbidities significantly increasing procedural risk. A new alternative procedure, balloon pulmonary angioplasty [BPA] has been proposed for patients with inoperable CTEPH or persistent pulmonary hypertension after pulmonary endarterectomy (PEA) and is currently characterized with good outcome in functional capacity, hemodynamic parameters, biomarkers, and health-related quality of life.

Exercise stress tests of the pulmonary circulation are used in workup and diagnosis of pulmonary hypertension as a hemodynamic abnormality. The approach has allowed identification of patients with normal or marginally increased mPAP at rest but with symptomatic increases in mPAP at exercise, related to either increased resistance or increased left atrial pressure. Although this differential diagnosis is of obvious therapeutic relevance, guidelines about exercise stress studies of the pulmonary circulation have not been developed until now for lack of robust evidence allowing for a consensus on clearly defined cutoff values.

Neither the pathophysiology of the exercise limitation nor the underlying mechanisms of the BPA - induced improvement were studied before. Therefore the aim of this study is to assess the hemodynamic effects of BPA treatment on the pressure-flow relationship in the pulmonary vasculature and the pulmonary vascular compliance. Furthermore, the investigators will explore possible differences in treatment effect across centers. Especially explore the timing of medical therapy vs balloon angioplasty.

.

ELIGIBILITY:
Inclusion Criteria:

-Patients with CTEPH or CTED eligible for balloon pulmonary angioplasty.

Exclusion Criteria:

-Patients unable to perform ergometer exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Slope of mPA/CO after BPA | 6 months after last BPA session
  Change from Baseline in Slope of mean pulmonary artery pressure/cardiac output after BPA at 6 months

SECONDARY OUTCOMES:
Change in resting PVR after BPA | 6 months after last BPA session
  Change from Baseline in pulmonary vascular resistance (PVR) after BPA at 6 months
Change in 6 MWT after BPA | 6 months after last BPA session
  Change from Baseline in 6 minute walk test (MWT) after BPA at 6 months
Change in NT-proBNP after BPA | 6 months after last BPA session
  Change from Baseline in NT-proBNP after BPA at 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Department of cardiology, Aarhus University Hospital, Aarhus, Denmark
- Nagoya University Hospital, Nagoya, Japan
- European Health Center, Otwock, Poland

IPD SHARING:
Plan to Share IPD: No